CLINICAL TRIAL: NCT00858325
Title: A Two Cohort, Open Label, Single and Multiple Dose Pharmacokinetic Study of 4mg/Kg and 6mg/Kg Doses of Daptomycin in Healthy Chinese Subjects Living in China
Brief Title: Pharmacokinetic Study of Daptomycin in Healthy Chinese Subjects Living in China
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Mathew Lo, Regional Product Director-Cubicin, AstraZeneca Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1790C00002
Record Dates: First submitted 2009-03-06; First posted 2009-03-09 (Estimated); Last update posted 2010-01-22 (Estimated); Status verified 2010-01

CONDITIONS: Healthy
Keywords: Cubicin; PK; China Registration; Pharmacokinetics
MeSH Terms: interventions — Daptomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Daptomycin — 4mg/kg and 6 mg/kg dissolved in 0.9% sodium chloride for injection, administered intravenously over 30 minutes.
  Other Names: Cubicin

SUMMARY:
The primary objective of this study is to characterise the pharmacokinetics and dose proportionality of daptomycin after single and multiple (once daily) 4mg/kg and 6 mg/kg doses of daptomycin in healthy Chinese volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Men or women (not of childbearing potential) of Chinese ethnicity
* Weight between 55Kg to 90Kg and have a Body Mass Index (BMI) between 18 and 25 kg/m2
* Have a calculated creatinine clearance within range from 80 to 120 ml/min inclusive

Exclusion Criteria:

* Unable to discontinue use of HMG-CoA reductase inhibitor therapy within 7 days prior to first dose of study drug through discharge from unit
* CPK > 2X ULN (upper limit of normal)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-02; Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic data will be obtained from the analysis of blood and urine samples that will be obtained at specific time points throughout the study. The pharmacokinetic samples will be collected on days 1, 4 through 8 and 9. | On therapy evaluation on Day1~9.

SECONDARY OUTCOMES:
Safety parameters (Incidence of AEs and SAEs, Deaths, Premature discontinuation due to an AE, regardless of relationship to study medication; Clinical lab data; Vital signs; ECG; Physical exam findings; Concomitant medications and adjunctive procedures). | On therapy evaluation on Day1~9.

CONTACTS AND LOCATIONS:
Overall Officials: Gang Chen, MD, Study Chair — AZ Pharmaceuticals - China; Haiyan Li, MD, Principal Investigator — Peking University Third Hospital
Locations (1):
- Research Site, Beijing, China